CLINICAL TRIAL: NCT04082650
Title: Vitamin D Supplementation Prior to in Vitro Fertilization in Women With Polycystic Ovary Syndrome: a Protocol of a Multicenter Randomised Double-blind Placebo-controlled Clinical Trial
Brief Title: Vitamin D and Pregnancy Outcome in PCOS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Principal Investigator, Dan Zhang, Vice president and Professor, Women's Hospital School Of Medicine Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VDPI
Record Dates: First submitted 2019-09-04; First posted 2019-09-09 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Polycystic Ovary Syndrome; in Vitro Fertilization
Keywords: Polycystic Ovary Syndrome; in vitro fertilization; Vitamin D; randomized trial
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and most researchers will be unaware of the actual grouping. Only two researchers who are not involved in participant management or data analysis will be aware of the grouping.
  Vitamin D and placebo pills with identical package, size, colour and appearance will be used in this trial. In general, there should be no need to unblind the allocation. If urgent unbinding to participants is necessary, the allocation will be disclosed to the treating physician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D (Experimental): Participants in the intervention group will be treated with vitamin D 4000IU (800IU per pill, take five pills once each day) per day for around 12 weeks (till the triggering day).
  Interventions: Drug: vitamin D
- Placebo (Placebo Comparator): Participants in the control group will be treated with equal amount of placebo tablets per day for the same duration.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: vitamin D — 4000IU per day
  Other Names: non
  Arms: Vitamin D
Other: Placebo — The same doses with vitamin D
  Arms: Placebo

SUMMARY:
This multicenter double-blinded placebo-controlled randomised trial aims to evaluate the effectiveness of vitamin D supplementation prior to IVF on the live birth rate in women with PCOS. Women with PCOS scheduled for IVF will be enrolled. Eligible participants will be randomised 1:1 to receive oral capsules of 4000IU vitamin D per day or placebo for around 12 weeks until the day of triggering.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is one of the leading causes of female infertility, affecting around 5% of women with a child-bearing age in China. Vitamin D insufficiency is common in women with PCOS and is associated with lower live birth rates in these women. However, evidence regarding the effectiveness of vitamin D treatment in women with PCOS is inconclusive. This multicenter double-blinded placebo-controlled randomised trial aims to evaluate the effectiveness of vitamin D supplementation prior to IVF on the live birth rate in women with PCOS.

The investigators plan to enroll women with PCOS scheduled for IVF. Eligible participants will be randomised 1:1 to receive oral capsules of 4000IU vitamin D per day or placebo for around 12 weeks until the day of triggering. All IVF procedures will be carried out following a routine method in each center. Women will be followed up until six months after randomisation for those who fail to get pregnant after the completion of the first embryo transfer or delivery for those who get pregnant after the first embryo transfer. The primary outcome is live birth after the first embryo transfer. Primary analysis will be by intention-to-treat analysis. The investigators plan to recruit 860 women to demonstrate women treated with vitamin D have a higher live birth rate than those treated with placebo (48% versus 38%), accounting for 10% loss to follow-up with a significance level at 0.05 and a power of 80%.

ELIGIBILITY:
Inclusion criteria

1. Women aged 20 to 42 years old;
2. Diagnosed with PCOS (Rotterdam Criteria);
3. Scheduled for IVF;
4. Written informed consent.

Exclusion criteria

1. Women who had three or more failed IVF cycles;
2. Women scheduled for preimplantation genetic testing;
3. Known Vitamin D allergy;
4. Women with a history of chronic absorption syndrome or bile dysplasia, or parathyroid dysfunction, or kidney stones, or blood Calcium ion concentration greater than 2.6mmol/L (normal value 2.25 - 2.75mmol/L (9 to 11mg/dl), or hyperphosphataemia (1.61mmol/L), or metabolic-related bone disease, or chronic diseases that may cause bone abnormalities (liver and kidney insufficiency);
5. Women receiving treatments for tuberculosis, convulsions, and epilepsy because medications treating these diseases may affect the metabolism of vitamin D.
6. Women undergoing an IVF treatment with donor oocytes.

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 876 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants with live birth | 1 day after delivery
  The primary outcome is live birth after the first embryo transfer. Live birth is defined as the delivery of at least one baby after 24 weeks of gestation that exhibits any sign of life.

SECONDARY OUTCOMES:
Number of Participants with Cumulative live birth | 6 months after randomization of the last participant
  Cumulative live birth: defined as live birth resulting from pregnancies that occur within 6 months after randomization.
Number of Participants with Clinical pregnancy | 4 weeks after embryo transfer
  Clinical pregnancy: defined as at least one gestational sac on ultrasound at around 7 weeks' gestation with the detection of heart beat activity after the completion of the first embryo transfer;
birth weight | The day of delivery
  Weight of newborns at delivery.
Number of Participants with miscarriage | 24 gestational weeks in maximum
  miscarriage was defined as a positive pregnancy test but no detectable heart rate before 24 weeks' gestation after the completion of the first transfer;
Number of Participants with Ongoing pregnancy | at 12 weeks' gestation
  defined as pregnancy with detectable heart rate at 12 weeks' gestation or beyond after the completion of the first transfer
Number of Participants with Biochemical pregnancy | 2 weeks after embryo transfer
  defined with a positive pregnancy test
Number of Participants with Ectopic pregnancy | 4 weeks after embryo transfer
  defined as embryo implanted at any site other than the endometrial lining of the uterus cavity after the completion of the first transfer
Number of Participants with Ovarian hyperstimulation syndrome | From the day of oocyte retrieval to two weeks after embryo transfer
  defined according to the Golan criteria. Moderate OHSS is diagnosed by the presence of ascites on ultrasonography in addition to abdominal distension and discomfort with or without nausea, vomiting and/or diarrhea. Severe OHSS is diagnosed when there is clinical evidence of ascites and/or hydrothorax or breathing difficulties with or without hemoconcentration, coagulation abnormalities and diminished renal function.
Number of available embryos for transfer | 5 days after oocyte retrieval
  non
Number of Participants with Pre-eclampsia | 20 weeks of gestation till delivery
  defined as the development of gestational hypertension with proteinuria (≥300 mg/24-hour urine collection or 30 mg/dL in single urine sample) of new onset after 20 weeks of gestation after the completion of the first transfer
Number of Participants with Gestational hypertension | 20 weeks of gestation till delivery
  defined as the development of blood pressure greater than 140/90 mmHg after pregnancy without proteinuria or other signs of preeclampsia after the completion of the first transfer;
Number of Participants with Premature rupture of membrane | The day of delivery
  PROM was defined as rupture of the amniotic membranes before the onset of labor including PROM at term and preterm PROM.
Number of Participants with Postpartum hemorrhage | 1 day after delivery
  defined as the loss of 500 ml of blood or more after completion of the third stage of labor after the completion of the first transfer
Number of Participants with Preterm delivery | 1 day after delivery
  Defined as delivery of a fetus at less than 37 and more than 28 weeks' gestational age after the completion of the first transfer
Number of Participants with Gestational diabetes mellitus | Up to ten months once the participants get pregnancy
  defined as carbohydrate intolerance of variable severity with onset or first recognition during pregnancy as determined from the diagnosis in the obstetrical medical record
Number of Participants with Placenta previa | after 24 weeks of gestation
  defined as a placenta that is implanted over or very close to the internal cervical orifice
Number of Participants with Stillbirth | 1 day after delivery
  defined as the absence of signs of life at or after birth after the completion of the first transfer
Apgar score | 1 minute or 5 minutes after delivery
  non
Serum Vitamin D binding protein, glucose, insulin, Calcium ion concentration | The day of oocyte retrieval
  non
Serum vitamin levels | One day before oocyte retrieval
  Serum vitamin levels at the triggering day

CONTACTS AND LOCATIONS:
Overall Officials: Dan Zhang, M.D. Ph.D., Principal Investigator — Women's Hospital School Of Medicine Zhejiang University
Locations (2):
- China (2):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Women's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
All data relevant to the study will be generated in the article or uploaded as supplementary information. Deidentified participant data will be available from Dr. Dan Zhang (zhangdan@zju.edu.cn) on a reasonable request. Protocols and statistical analysis plans will be included as supplementary information.

REFERENCES:
- [Derived] Hu KL, Gan K, Wang R, Li W, Wu Q, Zheng B, Zou L, Zhang S, Liu Y, Wu Y, Chen R, Cao W, Yang S, Liu FT, Tian L, Zeng H, Xu H, Qiu S, Yang L, Chen X, Pan X, Wu X, Mol BW, Li R, Zhang D. Vitamin D supplementation prior to in vitro fertilisation in women with polycystic ovary syndrome: a protocol of a multicentre randomised, double-blind, placebo-controlled clinical trial. BMJ Open. 2020 Dec 8;10(12):e041409. doi: 10.1136/bmjopen-2020-041409. PMID 33293396